CLINICAL TRIAL: NCT04506957
Title: Non-invasive Continuous Total Hemoglobin Measurement by Pulse CO-Oximetry in Major Spine Surgery
Brief Title: Non-invasive Continuous Total Hemoglobin Measurement by Pulse CO-Oximetry
Acronym: SpHb
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Klinik Hirslanden, Zurich (Other)
Responsible Party: Principal Investigator, Werner Baulig, Prof. Dr. med. Werner Baulig, Klinik Hirslanden, Zurich
Other Study IDs: Pulse-CO Oximetry Hemoglobin
Record Dates: First submitted 2020-08-07; First posted 2020-08-10 (Actual); Last update posted 2020-09-04 (Actual); Status verified 2020-09

CONDITIONS: Transcutaneous Continuous Hemoglobin Measurement

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: Pulse CO-Oximetry Hemoglobin measurement transcutaneous — this is an observational Investigation, in which transcutaneous continuous hemoglobin detection using Pulse-CO-Oximetry is compared with co-oximetrically measured Hemoglobin using a blood gas analyzer device
  Other Names: interventions are only performed based on co-oximetry hemoglobin measurement using a blood gas analyzer

SUMMARY:
This study is a data collection/sampling project for transcutaneous continuous Pulse CO-Oximetry and accessories (SW-Version Radical-7® Pulse CO-Oximeter with the Masimo rainbow SETTM, V1.6.2.4i Masimo Corp., Irvine, CA, USA, and the RD rainbow SET-2, Rev-O Fingersensor). The device received the CE Mark in 2012 and is approved by the Swiss Medic for clinical use. The Radical-7 device isolates multiple (7+) wavelengths of light of arterial signals using adaptive filters. It provides continuous noninvasive monitoring of arterial oxygen saturation (RadSpO2), pulse rate (RadPR), carboxyhaemoglobin saturation (SpCO), methaemoglobin saturation (SpMET), total haemoglobin concentration in g/dl (SpHb) and/or respiration rate (RRa). Additionally, Low Signal IQ (Low SIQ), Perfusion Index (PI), Pleth Variability Index (PVI), total arterial oxygen content (SpOC), Haematocrit (SpHCT), Signal identification Quality (SIQa), Respiration Indicator (RI) are displayed.The purpose of this prospective study is to investigate the reliability of non-invasive continuously measured SpHb by the Masimo Radical-7® Pulse co-oximeter (Radical 7 device) under steady state conditions by comparison against simultaneously invasive measured arterial haemoglobin concentrations (CoOxHb) in major spine surgery patients, in which high blood loss was expected

DETAILED DESCRIPTION:
The objective of this investigation is the comparison of CoOxHb, HCT and SaO2 values of a blood gas analyzer (ABL 825, Radiometer Medical A/S) with simultaneously measured SpHb values of the Radical 7 device during the procedure of major spine surgery.

The primary endpoint of the study is the reliability of SpHb to detect CoOxHb and its changes during the process Secondary endpoint is the reliability of RadSpO2, RadPR, SpHCT and SpMET to detect SaO2, PR, HCT and MetHb and its changes during the process.

Inclusion criteria:

1. Patients scheduled for major spine surger
2. Age 18 years and older
3. Written consent of the participation after clarification about the study

Exclusion criteria:

1. No consent to participate
2. No German comprehension
3. Black skin patients
4. Patients with COVID-19 illness All patients were monitored based on the institutional routine monitoring for major spine surgery (continuous 2-channel electrocardiogram, a continuous invasive arterial blood pressure monitoring via fluid-filled cather system, inserted in the radial artery mainly of the non-dominant hand, SpO2, and in the case of high-risk patient a triple-lumen central venous line). Then a single use finger sensor (MasimoSet RD rainbow SET SpHb SpMet-Sensor) is attahed to the ring finger of the hand, where the catheter is introduced in the radial artery.

During the surgery routinely, arterial blood samples are drawn before induction of Anaesthesia, every 45 min and after acute blood loss during surgery. With each blood sample for a blood gas analysis the SpHb, SpMet, PI, PVI and the low SQI are recorded.

No additional blood sampling is necessary to perfom this investigation

50 patients will be included and the duration of the study is 24 month's Sample size calculation was performed with the StatsDirect Statistical Software Version 2.8.0 2013 (StatsDirect Ltd, Altrincham, UK) and revealed a sample size of 95 paired SpHb and CoOxHb measurements to achieve a power of 0.9, α = 0.05 to detect a mean difference (bias) of CoOxHb and SpHb of 0.50 g/dl with an estimated standard deviation (SD) of 1.0g/dl. The mean difference is determined based on previous investigations. Continuous variables are tested for normal distribution with the Kolmogorov-Smirnow test. Normally distributed data are expressed as mean ± standard deviation (SD); median, interquartile range (IQR ; 25th to 75th percentile) and [maximum] are specified when the data were not normally distributed. Categorical variables are presented as number and percentage (%). For subgroup analysis continuous variables are compared using the t-test or Mann-Whitney U test, when appropriate. All tests are two-sided and a P-value < 0.05 was determined to be significant.

For all determinants that might have an impact on the fault detection of the SpHb stepwise multiple regressions analysis was performed. Correlation is evaluated by Spearman rank test. To determine agreement of the methods, the Bland Altman analysis for repeated measurements is performed for SpHb and CoOcHb.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for major spine surgery
* Written consent of the participation after clarification about the study

Exclusion Criteria:

1. No consent to participate
2. No German comprehension
3. Black skin patients
4. Patients with COVID-19 illness

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for major spine surgery
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-12-01 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Reliability of SpHb to detect CoOxHb and its changes | 24 months
  Co-oximetry hemoglobin values from blood gas analyzer is simultaneous compared with the transcutaneous detected SpHb (Pulse CO-Oximetry hemoglobin measurement). Linear correlation and Bland Altman Analysis are performed for analysis these data pairs

CONTACTS AND LOCATIONS:
Overall Officials: Werner Baulig, MD, Principal Investigator — Klinik Im Park

IPD SHARING:
Plan to Share IPD: No
it is not planned to make individual participant data available to other researchers

REFERENCES:
- [Background] Baulig W, Seifert B, Spahn DR, Theusinger OM. Accuracy of non-invasive continuous total hemoglobin measurement by Pulse CO-Oximetry in severe traumatized and surgical bleeding patients. J Clin Monit Comput. 2017 Feb;31(1):177-185. doi: 10.1007/s10877-015-9816-2. Epub 2015 Dec 19. PMID 26686689